CLINICAL TRIAL: NCT00994279
Title: Yoga or Wellness Education During Breast Cancer Treatment: Establishing Community-Based Partnerships
Brief Title: Yoga or Educational Wellness Class for Women With Stage I, Stage II, or Stage III Breast Cancer Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00011383; U10CA081851 (NIH); REBACCCWFU97309 (Other: NCI)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Depression; Fatigue; Sleep Disorders
Keywords: fatigue; depression; sleep disorders; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Sleep Wake Disorders | interventions — Yoga; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Yoga Intervention (Active Comparator): Yoga Intervention
  Interventions: Behavioral: Yoga
- Arm 2: Educational Wellness Group (Active Comparator): Educational Wellness Group
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Yoga — Yoga sessions
  Arms: Arm 1: Yoga Intervention
Behavioral: Education — Educational Wellness Group
  Arms: Arm 2: Educational Wellness Group

SUMMARY:
RATIONALE: Yoga and wellness classes may reduce fatigue and improve mood, sleep, and quality of life in women receiving chemotherapy for breast cancer. It is not yet known whether yoga is more effective than wellness education for women with breast cancer who are undergoing chemotherapy.

PURPOSE: This randomized phase II trial is studying a community-based yoga class to see how well it works compared with an educational wellness class for women with stage I, stage II, or stage III breast cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the participation rate, accrual, adherence, and retention to a community-based study of yoga vs an active control (wellness education) in women with stage I-III breast cancer undergoing chemotherapy.

Secondary

* To obtain estimates of the variability of women's self-reported fatigue and depressive symptoms, sleep quality, and health-related quality of life from baseline to the end of the intervention at 10 weeks.
* To obtain estimates of the efficacy of a community-based yoga intervention in women with breast cancer.
* To standardize the yoga protocol for use in multiple community settings with breast cancer patients, and ascertain that yoga teachers can adhere to a uniform protocol.

OUTLINE: This is a multicenter study. Patients are stratified according to CCOP site and chemotherapy-treatment status (planning vs started). Patients are randomized to 1 of 2 intervention arms.

Patients must begin their class or group within 3 weeks of starting chemotherapy. All women enter their class or group on a rolling basis so that their class or group coincides with the weeks that they receive chemotherapy treatments.

* Arm I (Yoga intervention): In weeks 1-10, patients attend a community-based weekly 75-minute Integral Yoga class led by an experienced yoga teacher specifically trained in adapting yoga for people with cancer. The yoga class includes postures, deep relaxation, breathing practices, and meditation to create a profound experience of peace and well-being. Women are asked to attend ≥ 8 of 10 classes over a 12-week period to allow for missed classes. Women are also provided with a yoga mat, associated yoga props (bolster, strap), and a 45-minute cancer-specific yoga DVD for home practice. Women are asked to practice yoga outside of the class at least twice per week, and are encouraged to practice more frequently than that.
* Arm II (Active control): Patients meet for a weekly 75-minute wellness education group in weeks 1-10 (women may make-up missed classes during weeks 11 and 12). The group focuses on issues that women with breast cancer face as they undergo treatment; topics include symptom management, financial and insurance issues, emotional issues/coping with cancer, communicating with healthcare providers/navigating the healthcare system, healthful eating/cooking demonstrations, sexual issues/fertility/body image, mobilizing social support/impact of cancer on family and friends, survivorship (advocacy) opportunities, and common concerns/fear of recurrence. Women are provided with reading materials relevant to the topics that will be covered in each group meeting and are asked to spend approximately 45 minutes twice weekly reading these materials and incorporating any relevant principles/ideas into their daily lives. Women may request additional reading materials in further topics of interest from the group facilitators.

Patients complete questionnaires at baseline and at weeks 5, 10, and 14 to assess fatigue (FACIT-Fatigue), depressive symptoms (Center for Epidemiologic Studies-Depression Scale [CES-D]), treatment-related symptoms (M.D. Anderson Symptom Inventory [MDASI]), sleep disturbance (Medical Outcomes Study Sleep Measure [MOS-Sleep]), and health-related quality of life (Functional Assessment of Cancer Therapy-Breast [FACT-B]). Patients also track time spent on all home-yoga practice (arm I) or wellness-group homework (arm II). After the intervention (week 10), patients are asked to provide feedback on the program. Yoga/Wellness teachers will completion intervention feedback forms 6 months from the start of the first intervention and at completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Women will be eligible if they are:

* Scheduled to begin chemotherapy treatment within 3 weeks of study registration, or able to start Yoga/Wellness sessions prior to second chemotherapy treatment.
* ≥18 years of age.
* Physically able to attend yoga classes (simply meaning that they can physically make it to the intervention session and are able to sit on a chair or lie on the floor) (ECOG Performance Status rating 0-2; Zubrod et al., 1960).
* Diagnosed with breast cancer Stages I-III.
* Chemotherapy is anticipated to continue during the 10 weeks of the study intervention.
* 2-8 weeks post-completion of breast surgery (unless receiving neoadjuvant chemotherapy).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Have practiced yoga on a regular basis (at least once a week) within the past 4 weeks to recruit women who are not already regularly practicing yoga. Given that the benefits of yoga are likely more immediate than long-term, however, we will enroll women who have previously had a yoga practice.
* Are being treated with surgery and/or radiation therapy and/or hormonal treatment only and/or Herceptin therapy only (no chemotherapy).
* Anticipate undergoing surgery related to their breast cancer or receipt of radiation therapy during the study period.
* Have regularly engaged in moderate (activity that makes you breathe somewhat harder than normal; may include carrying light loads, bicycling at a regular pace, fast walking, tennis, easy swimming, or popular or folk dancing) or vigorous (activity that causes heavy breathing, sweating, rapid fatigue; it can only be sustained for very short periods of time, like running or swimming strongly) physical activity at least 3-5 days per week (on average) within the past 4 weeks.

Pregnant women will not be excluded from this study because the study intervention(s) pose no risk of potential for teratogenic or abortifacient effects. In fact, gentle yoga practice is quite safe for pregnant women and poses can be slightly modified, if needed. The anticipated number of pregnant women eligible to enroll is minimal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-10-14 (Actual); Study Completion 2011-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three NCI CCOP sites between 1/2010 and 8/2011
Period: Overall Study
Arm/Group | Arm 1: Yoga Intervention | Arm 2: Educational Wellness Group
Started | 22 | 18
Completed | 18 | 13
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Toxicity | 1 | 0
Not completed — Multiple reasons | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Yoga Intervention | Arm 2: Educational Wellness Group | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 50 [29 to 83] | 45 [29 to 64] | 47 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Proportion of participants completing the 10 week study
Time Frame: 10 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Yoga Intervention | Arm 2: Educational Wellness Group
Number analyzed (Participants) | 22 | 18
percentage of participants | 82 [60 to 95] | 89 [65 to 99]
Statistical Analysis 1: Comparison: Arm 1: Yoga Intervention vs Arm 2: Educational Wellness Group; Null hypothesis is that the two arms will not differ in retention at 14 weeks; Test type: Superiority or Other; p = .53, Chi-squared

2. Secondary Outcome: Fatigue at 10 Weeks
Description: FACIT-Fatigue patient reported outcome. This questionnaire consists of 13 questions answered on a 0 to 4 scale with a min of 0 and a max of 52. Higher scores indicate less fatigue.
Time Frame: 10 weeks
Population: Participants with 10 week outcome data. Note that one participant in the Wellness group was missing this outcome even though they completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Yoga Intervention | Arm 2: Educational Wellness Group
Number analyzed (Participants) | 18 | 15
units on a scale | 30.2 (2.6) | 30.1 (2.9)
Statistical Analysis 1: Comparison: Arm 1: Yoga Intervention vs Arm 2: Educational Wellness Group; Null hypothesis is that the two groups would not differ in fatigue at 10 weeks; Test type: Superiority or Other; p = .98, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Sample includes all patients with follow-up toxicity assessments. This number is different from the sample size in other analyses because some participants provided follow-up toxicity assessments before they went off study. Patients were asked about adverse events at each assessment visit.
Arm/Group | Arm 1: Yoga Intervention | Arm 2: Educational Wellness Group
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/17
Other Adverse Events (participants affected / at risk) | 11/21 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Yoga Intervention (N=21) | Arm 2: Educational Wellness Group (N=17)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Yoga Intervention (N=21) | Arm 2: Educational Wellness Group (N=17)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 3 (6) | 2 (4)
Infections and Infestations (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1)
Musculoskeletal/Soft tissue = Cartilage Tears (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (General disorders) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in Extremity (Nervous system disorders) | 8 (12) | 4 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes